CLINICAL TRIAL: NCT05629611
Title: Efficacy and Safety Evaluation of Advanced Vessel Sealing Device (Vi-sealer)
Brief Title: Efficacy and Safety Evaluation of Vi-sealer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hyun Park (Other)
Responsible Party: Sponsor-Investigator, Hyun Park, Professor, CHA University
Organization: CHA University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KGOG4009_Vi-TLH
Record Dates: First submitted 2022-10-31; First posted 2022-11-29 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Benign Gynecologic Neoplasm
Keywords: Advanced hemostatic devices; Advanced energy devices; Ligasure; Laparoscopic total hysterectomy; Vi-sealer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Study 1 Vi-Sealer (Experimental): This group of women undergoing hysterectomy is randomized to the energy device, Vi-sealer.
  Interventions: Device: Vi-Sealer
- Study 1 Ligasure (Active Comparator): This group of women undergoing hysterectomy is randomized to the energy device, Ligasure.
  Interventions: Device: Ligasure
- Study 2 Vi-sealer (Experimental): This group of women undergoing hysterectomy is randomized to the energy device, Vi-sealer.
  Interventions: Device: Vi-Sealer
- Study 2 Other AHD (Active Comparator): This group of women undergoing hysterectomy is randomized to energy devices other than Ligasure.
  Interventions: Device: Other AHD

INTERVENTIONS:
Device: Vi-Sealer — using Reusable device, Vi-Sealer
  Arms: Study 1 Vi-Sealer; Study 2 Vi-sealer
Device: Ligasure — using Ligasure
  Arms: Study 1 Ligasure
Device: Other AHD — Using other AHDs such as Thunderbeat, Harmonic scalpel, Caiman®, Enseal, etc. except Ligasure
  Arms: Study 2 Other AHD

SUMMARY:
This study's primary goal is to compare the efficacy and safety of the novel advanced hemostatic device(AHD), Vi-Sealer, with conventional AHDs in laparoscopic total hysterectomy for patients with benign gynecologic neoplasm.

DETAILED DESCRIPTION:
Vi-Sealer is a reusable advanced bipolar electrode with an interchangeable blade. This study evaluates the efficacy and safety of the Vi-Sealer by comparing it with other advanced hemostatic devices, such as Ligasure, Enseal, Thunderbeat, Harmonic scalpel, etc. The economic evaluation of the device compared with other disposable devices would also be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20 to 65 years
2. Clinically diagnosed with benign gynecologic neoplasms (eg. adenomyosis, uterine fibroids, etc.)
3. Eligible for hysterectomy
4. Signing an written consent form indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study prior to any other study-related assessments or procedure

Exclusion Criteria:

1. Large uterus size over 16 weeks of gestational age
2. Cervical or intraligamentary fibroids
3. Severe endometriosis (stage 3 or 4)
4. Suspected malignancy of the uterus or adnexa
5. Contraindicated for the use of energy devices (such as implantable cardioverter defibrillators, pacemakers)
6. Previous pelvic surgery ≥ 3 times
7. Not suitable for laparoscopic surgery

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Operative procedure time | through study completion, an average of 1 year
  Measure the time consumed from the initial skin incision to the closure of abdominal trocar sites
Estimated blood loss | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Estimated medical cost of device | within 6 weeks after intervention
  Medical costs according to hemostatic instrument use
Device evaluation score | through study completion, an average of 1 year
  Ergonomics and subjective hemostatic performances assessed by surgeons using the survey
Adverse events | within 6 weeks after intervention
  Collect only for adverse events that have a relationship with medical devices for clinical trials

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong C, Goh A, Merkur H. Comparison of surgical outcomes using Gyrus PKS vs LigaSure in total laparoscopic hysterectomy: A randomised controlled trial. Aust N Z J Obstet Gynaecol. 2020 Oct;60(5):790-796. doi: 10.1111/ajo.13217. Epub 2020 Jul 29. PMID 32729141
- [Background] Holloran-Schwartz MB, Gavard JA, Martin JC, Blaskiewicz RJ, Yeung PP Jr. Single-Use Energy Sources and Operating Room Time for Laparoscopic Hysterectomy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2016 Jan;23(1):72-7. doi: 10.1016/j.jmig.2015.08.881. Epub 2015 Aug 28. PMID 26318400
- [Background] Janssen PF, Brolmann HA, van Kesteren PJ, Bongers MY, Thurkow AL, Heymans MW, Huirne JA. Perioperative outcomes using LigaSure compared with conventional bipolar instruments in laparoscopic hysterectomy: a randomised controlled trial. BJOG. 2011 Dec;118(13):1568-75. doi: 10.1111/j.1471-0528.2011.03089.x. Epub 2011 Sep 6. PMID 21895949
- [Background] Hasanov M, Denschlag D, Seemann E, Gitsch G, Woll J, Klar M. Bipolar vessel-sealing devices in laparoscopic hysterectomies: a multicenter randomized controlled clinical trial. Arch Gynecol Obstet. 2018 Feb;297(2):409-414. doi: 10.1007/s00404-017-4599-y. Epub 2017 Dec 8. PMID 29222641
- [Background] Winter ML, Mendelsohn SA. Total laparoscopic hysterectomy using the harmonic scalpel. JSLS. 1999 Jul-Sep;3(3):185-6. PMID 10527328
- [Background] Shiber LJ, Ginn DN, Jan A, Gaskins JT, Biscette SM, Pasic R. Comparison of Industry-Leading Energy Devices for Use in Gynecologic Laparoscopy: Articulating ENSEAL versus LigaSure Energy Devices. J Minim Invasive Gynecol. 2018 Mar-Apr;25(3):467-473.e1. doi: 10.1016/j.jmig.2017.10.006. Epub 2017 Oct 12. PMID 29032252
- [Background] Rothmund R, Kraemer B, Brucker S, Taran FA, Wallwiener M, Zubke A, Wallwiener D, Zubke W. Laparoscopic supracervical hysterectomy using EnSeal vs standard bipolar coagulation technique: randomized controlled trial. J Minim Invasive Gynecol. 2013 Sep-Oct;20(5):661-6. doi: 10.1016/j.jmig.2013.04.014. Epub 2013 Jun 20. PMID 23791399
- [Background] Lee CL, Wu KY, Huang CY, Yen CF. Comparison of LigaSure tissue fusion system and a conventional bipolar device in hysterectomy via natural orifice transluminal endoscopic surgery (NOTES): A randomized controlled trial. Taiwan J Obstet Gynecol. 2019 Jan;58(1):128-132. doi: 10.1016/j.tjog.2018.11.024. PMID 30638466
- [Background] Honeck P, Wendt-Nordahl G, Bolenz C, Peters T, Weiss C, Alken P, Michel MS, Hacker A. Hemostatic properties of four devices for partial nephrectomy: a comparative ex vivo study. J Endourol. 2008 May;22(5):1071-6. doi: 10.1089/end.2007.0236. PMID 18429683
- [Background] Landman J, Kerbl K, Rehman J, Andreoni C, Humphrey PA, Collyer W, Olweny E, Sundaram C, Clayman RV. Evaluation of a vessel sealing system, bipolar electrosurgery, harmonic scalpel, titanium clips, endoscopic gastrointestinal anastomosis vascular staples and sutures for arterial and venous ligation in a porcine model. J Urol. 2003 Feb;169(2):697-700. doi: 10.1097/01.ju.0000045160.87700.32. PMID 12544345
- [Background] Timm RW, Asher RM, Tellio KR, Welling AL, Clymer JW, Amaral JF. Sealing vessels up to 7 mm in diameter solely with ultrasonic technology. Med Devices (Auckl). 2014 Jul 30;7:263-71. doi: 10.2147/MDER.S66848. eCollection 2014. PMID 25114600
- [Background] Nieboer TE, Steller CJ, Hinoul P, Maxson AJ, Schwiers ML, Miller CE, Coppus SF, Kent AS. Clinical utility of a novel ultrasonic vessel sealing device in transecting and sealing large vessels during laparoscopic hysterectomy using advanced hemostasis mode. Eur J Obstet Gynecol Reprod Biol. 2016 Jun;201:135-9. doi: 10.1016/j.ejogrb.2016.03.035. Epub 2016 Apr 14. PMID 27124666
- [Background] Sandberg EM, la Chapelle CF, van den Tweel MM, Schoones JW, Jansen FW. Laparoendoscopic single-site surgery versus conventional laparoscopy for hysterectomy: a systematic review and meta-analysis. Arch Gynecol Obstet. 2017 May;295(5):1089-1103. doi: 10.1007/s00404-017-4323-y. Epub 2017 Mar 29. PMID 28357561
- [Background] Park JY, Nho J, Cho IJ, Park Y, Kim DY, Suh DS, Kim JH, Nam JH. Laparoendoscopic single-site versus conventional laparoscopic-assisted vaginal hysterectomy for benign or pre-invasive uterine disease. Surg Endosc. 2015 Apr;29(4):890-7. doi: 10.1007/s00464-014-3747-8. Epub 2014 Aug 9. PMID 25106721
- [Derived] Kim M, Seong SJ, Kim K, Kim SW, Park ST, Kim WY, Choi YJ, Hong DG, Park H. Efficacy and safety evaluation of a reusable advanced hemostatic device (Vi-Sealer) during total laparoscopic hysterectomy in South Korea (KGOG4009/Vi-TLH trial): study protocol for a multicenter, open-label, non-inferiority randomized controlled trial. Trials. 2025 Nov 7;26(1):480. doi: 10.1186/s13063-025-09222-w. PMID 41204237